CLINICAL TRIAL: NCT06314360
Title: Comparison of Foot Posture, Plantar Pressure, and Postural Balance in Individuals With Patellofemoral Pain and Healthy Individuals
Brief Title: Comparison of Foot Posture, Plantar Pressure, and Postural Balance in Patellofemoral Pain Patients and Healthy Subjects
Status: Enrolling by invitation | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, HANDE GUNEY, Principal Investigator, Head of Early Orthopaedic Rehabilitation Unit, Hacettepe University
Other Study IDs: BAP_PFS
Record Dates: First submitted 2024-01-26; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: patellofemoral pain; pedobarography; postural stability; foot posture; functionality
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with Patellofemoral Pain: Demographic data, pain information, limb dominancy will be collected. Then, functional status will be assessed with Kujala Patellofemoral Pain Form; foot posture will be evaluated with Foot Posture Index; plantar pressure and postural balance values will be collected with the K-Invent K-Plates device.
  Interventions: Other: No intervention.
- Healthy Control Subjects: Demographic data, limb dominancy will be collected. Then, functional status will be assessed with Kujala Patellofemoral Pain Form; foot posture will be evaluated with Foot Posture Index; plantar pressure and postural balance values will be collected with the K-Invent K-Plates device.
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — There is no intervention in this study.

SUMMARY:
Patellofemoral pain syndrome (PFS) is a musculoskeletal problem characterized by pain felt in the front of the knee or behind the patella, commonly affecting individuals in adolescence or young adulthood, especially those engaged in sports such as cycling and running. It is one of the most encountered knee injuries and can have a poor prognosis. The intensity of knee pain increases during functional activities such as stair climbing, squatting, running, and jumping due to the increased patellofemoral joint reaction force.

A disturbance in postural stability is observed in individuals with PFS due to pain during functional activities. Studies examining changes in foot posture, plantar pressure, and postural balance in individuals with PFS are quite limited and controversial. Moreover, research that simultaneously investigates these parameters and interprets the results is scarce. Some studies have utilized detailed technical systems such as medical imaging or motion analysis, while practical methods incorporating foot posture and plantar pressure analyses are available and easy to use in clinical settings.

There is a lack of literature on the easy assessment and interpretation of plantar pressure, postural balance, and functional activities in individuals with PFS. Within the scope of this project, the plan is to assess plantar pressure, postural balance, and functional activities in individuals with PFS. The aim is to quickly interpret the biomechanical changes occurring in these individuals and guide rehabilitation programs based on the obtained data.

The use of practical and fast assessment methods in planning treatments for PFS is crucial for early rehabilitation planning. Practical methods such as foot posture, plantar pressure, and postural balance assessments, which can be used in clinical settings, may provide benefits in shaping rehabilitation goals related to lower extremity alignment in individuals with PFS. The objective of this study is to compare the foot posture, plantar pressure, and postural stability of individuals with PFS with healthy individuals. Additionally, the investigators aim to investigate the relationship between foot posture, plantar pressure parameters, postural balance, and functional level in individuals with PFS. Through these objectives, it will be possible to identify potential parameters that could be effective in rehabilitation processes and contribute to determining treatment programs by revealing biomechanical changes in individuals with PFS.

DETAILED DESCRIPTION:
PFS, commonly referred to as pain felt in the front or behind the kneecap, is a prevalent lower extremity problem. It most commonly affects adolescents and young adults, especially those engaged in sports such as cycling and running. Although its etiology is not fully explained, factors such as increased load on anatomical structures, repetitive movements with excessive degrees of knee flexion, patellofemoral malalignment, and muscle strength losses contribute to the pain. PFS is a frequently encountered musculoskeletal problem that adversely affects the quality of life and functional status in young adults.

Changes in lower extremity alignment (dynamic valgus, varus, tibial rotation, etc.) and alterations in foot position (increased pronation posture) are among the most important factors leading to PFS. Increased foot pronation during ground contact in walking and in static standing is suggested to trigger the development of PFS. Studies have shown that increased force and pressure distribution in the medial forefoot, midfoot, and heel after long-distance runs are associated with PFS. Conversely, there are studies suggesting no difference in foot posture between individuals with PFS and healthy individuals. One method that can be preferred to assess foot posture (in static or dynamic positions) is the measurement of plantar pressure distribution. This measurement method, based on plantar pressure distribution, is described as a safe and non-invasive method that allows the examination of changes related to the locomotor system, especially foot biomechanics. There are also systems that assess foot pressure distribution concurrently with evaluating foot position. Studies in the literature have demonstrated an association between foot pronation and increased plantar pressure in the medial foot in individuals with PFS. Additionally, there are studies indicating that the distribution of plantar pressure is similar between individuals with PFS and healthy individuals or that foot pronation is less in individuals with PFS compared to healthy individuals. Therefore, a clear conclusion in the literature regarding the foot plantar pressure in individuals with PFS has not yet been reached.

The severity of pain in PFS increases not only during daily life activities such as climbing stairs, squatting, and standing up from sitting but also during sports activities such as running and jumping. Studies show that during activities where weight is transferred to a single extremity, such as single-leg squatting, individuals with PFS experience decreased hip flexion, increased hip adduction and internal rotation, and disrupted pelvic alignment. It is suggested that if pelvic alignment cannot be maintained during weight transfer, postural balance will be negatively affected. The number of studies examining postural balance in individuals with PFS is limited, and a consensus has not been reached.

The evaluation methods used in the aforementioned studies generally rely on radiological imaging or motion analysis systems. Only a limited number of studies have utilized foot posture assessment and plantar pressure analysis. The different assessment methods used make it difficult to draw clear relationships between the results. Therefore, there is a need for a comprehensive study that evaluates parameters such as foot posture, plantar pressure, postural balance, and functional status together in individuals with PFS.

The use of practical and fast assessment methods is crucial in planning treatments for PFS to enable early rehabilitation planning. Therefore, practical methods such as foot posture, plantar pressure distribution, and postural balance assessments, which can be used in clinical settings, may provide benefits in shaping rehabilitation goals related to lower extremity alignment in individuals with PFS. The aim of this study is to compare the foot posture, plantar pressure distribution, and postural balance parameters of individuals with PFS with healthy individuals and to investigate the relationship between these parameters in individuals with PFS.

ELIGIBILITY:
Inclusion criteria for individuals with PFS:

* Those who have been experiencing pain for at least 6 months
* Those who met the numerical pain criteria, defined as a minimum of 3 out of 10 points
* Having pain in the activities specifically identified as painful for PFP patients, including prolonged sitting, descending and ascending stairs/slopes, squatting, running, and jumping.

Inclusion criteria for healthy individuals:

* Those who are without any complaints related to the lower extremities in the last 6 months
* Those who have not undergone lower extremity surgery for any reason
* Those who do not have a diagnosis of neurological or orthopedic diseases

Exclusion criteria for individuals with PFS:

* Those with a history of lower extremity injury in the last 6 months
* Those who had patellofemoral dislocation and/or subluxation
* Those with meniscus and ligament lesions, bone anomalies
* Those who have undergone surgery on any lower extremity joint (hip, knee, or ankle)

Exclusion criteria for healthy individuals:

* Those with a history of lower extremity injury in the last 6 months
* Those who are asymptomatic with a history of patellofemoral dislocation and/or subluxation
* Those who are asymptomatic with meniscus and ligament lesions, bone anomalies
* Those who have undergone lower extremity surgery

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects who are diagnosed with patellofemoral pain syndrome, and healthy subjects.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Plantar Pressure | 3 minutes, in the baseline assessment session.
  Plantar pressure assessment will be performed with K-Invent K-Plates device. This device has two separate platforms measuring 320x160 mm. Participants will stand on the device with each foot on a platform and pressure data will be collected as max kg and weigth distribution.
Postural Stability | 20 minutes, in the baseline assessment session.
  Postural stability assessment will be performed with K-Invent K-Plates device. This device has two separate platforms measuring 320x160 mm. While the participants are on the device with each foot on a platform, bipodal and then unipodal stance data will be collected respectively. Data will be collected three times for 50 seconds for each stance and stability data such as center of pressure, velocity and ellipse area will be recorded. Higher values show poor balance scores.
Foot posture | 5 minutes, in the baseline assessment session.
  Foot Posture Index will be used to evaluate foot posture. FPI is a six-item clinical assessment tool used to evaluate foot posture. The six criteria used in the evaluation are talar head palpation, supra malleolar and infra malleolar curvature, position of the calcaneal in the frontal plane, protrusion in the talonavicular joint region, compliance of the medial longitudinal arch, and abduction/adduction of the forefoot. Each API component is scored from -2 to +2, with -2 representing clear signs of supination and +2 indicating positive signs of pronation. The total score ranges from -12 to +12. Total scores between 0 and +5 indicate normal/neutral foot posture. Values ≥ +6 are considered pronated foot, while values below 0 are considered supinated foot.
Functionality | 3 minutes, in the baseline assessment session.
  Functional status will be assessed using Kujala Patellofemoral Pain Form. The questionnare consists of 13 questions. These questions ask whether there is pain during going up and down stairs, squatting, running, jumping and sitting for long periods with the knees flexed; It evaluates whether there is limp, swelling or subluxation of the patella, the amount of atrophy in the quadriceps muscle, flexion deficit and the need for a walking aid. The scoring system ranges from 0-100 points, from worst to best.

SECONDARY OUTCOMES:
Pain Assessment | 1 minute, in the baseline assessment session.
  Pain will be evaluated using Numeric Analogue Scale. In this scale, the intensity of pain at the time of questioning will be recorded by the person choosing the value corresponding to the relevant number on a 10 cm long line shown between 0 (no pain) and 10 (unbearable pain). Two separate inquiries will be made, including pain at rest and during activity.
Limb dominance | 30 seconds, in the baseline assessment session.
  Limb dominance will be recorded by asking "Which leg do you prefer to kick a ball?". The answer to this question will be recorded as the dominant leg.

CONTACTS AND LOCATIONS:
Overall Officials: Hande Guney, Principal Investigator — Hacettepe University Faculty of Physical Therapy and Rehabilitation
Locations (1):
- Hacettepe University, Ankara, Ankara/Sıhhıye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No